CLINICAL TRIAL: NCT00003000
Title: Peripheral Effects of Opioid Analgesia in Patients Undergoing Axillary Node Dissection
Brief Title: Morphine for the Treatment of Pain in Patients With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Dr. Oscar Deleon, Roswell Park Cancer Institute
Other Study IDs: CDR0000065555; RPCI-DS-92-13
Record Dates: First submitted 1999-11-01; First posted 2004-07-30 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Pain
Keywords: pain
MeSH Terms: conditions — Pain | interventions — Fentanyl; Morphine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fentanyl citrate
Drug: morphine sulfate

SUMMARY:
RATIONALE: Morphine helps to relieve the pain associated with cancer surgery. Giving morphine in different ways may offer more pain relief.

PURPOSE: This randomized clinical trial is studying how well morphine injected directly into the underarm area works compared with morphine injected into the back of the shoulder in treating pain in patients who have breast cancer and who are undergoing axillary lymph node dissection.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether morphine injected at the site of surgery can control pain from surgery.

OUTLINE: This is a prospective, double blind, randomized study. Patients are randomized into 3 groups with 6 patients in each group. Group 1 receives morphine diluted in normal saline (NS), which is administered in the axillary region at the completion of surgery before surgical closure. The area is flooded and the solution is allowed to remain in the wound for 5 minutes. Group 2 (control group) receives NS only, administered in the same fashion as group 1. Group 3 receives morphine subcutaneously in the deltoid area, ipsilateral to the site of surgery, at the beginning of wound closure. Postoperatively, patients self-administer IV fentanyl analgesia through a patient controlled analgesia pump. Comparisons of daily IV fentanyl utilization is done among the three groups. Quality of pain is assessed via visual analog pain scores four times a day at 2, 4, 6, and 24 hours postoperatively.

PROJECTED ACCRUAL: A total of 18 patients will be accrued over a period of 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Patients with breast cancer who are scheduled to undergo axillary node dissection

PATIENT CHARACTERISTICS: See General Eligibility Criteria

PRIOR CONCURRENT THERAPY: No oral-equivalent doses of morphine greater than 10 mg a day -- Patient Characteristics-- Age: Not specified Sex: Not specified Other: Not allergic to morphine

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Breast Cancer Patients
Sampling Method: Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 1992-05; Primary Completion 2001-01 (Actual); Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States